CLINICAL TRIAL: NCT04654988
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Immunosuppression in Biopsy-proven Virus Negative Myocarditis or Inflammatory Cardiomyopathy
Brief Title: Study to Evaluate the Efficacy of Immunosuppression in Myocarditis or Inflammatory Cardiomyopathy.
Acronym: IMPROVE-MC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREDAZA/WUM/10-09-2020; 2020-003877-23 (EudraCT Number)
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: Myocarditis; Heart Failure; Endomyocardial Biopsy; Cardiomyopathies, Secondary; Immunosuppression
Keywords: myocarditis, cardiomyopathy, immunosuppression, biopsy
MeSH Terms: conditions — Myocarditis; Heart Failure; Cardiomyopathies | interventions — Prednisone; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppression (Experimental): Prednisone: 1 mg/kg daily for 4 weeks followed by gradually tapered dose for 5 months and Azathioprine: 2 mg/kg daily for 12 months
  Interventions: Drug: Prednisone; Drug: Azathioprine
- Placebo (Placebo Comparator): placebo matching prednisone: 1 mg/kg daily for 4 weeks followed by gradually tapered dose for 5 months and placebo matching azathioprine: 2 mg/kg daily for 12 months
  Interventions: Drug: Placebo Prednisone; Drug: Placebo Azathioprine

INTERVENTIONS:
Drug: Prednisone — Prednisone: 1 mg/kg daily for 4 weeks followed by gradually tapered dose for 5 months
  Arms: Immunosuppression
Drug: Azathioprine — Azathioprine: 2 mg/kg daily for 12 months
  Arms: Immunosuppression
Drug: Placebo Prednisone — Placebo Prednisone
  Arms: Placebo
Drug: Placebo Azathioprine — Placebo Azathioprine
  Arms: Placebo

SUMMARY:
Myocarditis can result in numerous complications, but there is paucity of data regarding optimal therapy, short- and long-term effects of possibly effective immunosuppressive therapy. The IMPROVE-MC study will provide high-quality scientific data about efficacy and safety of immunosuppressive therapy, non-invasive (MRI, biomarkers) and invasive diagnostics tests (endomyocardial biopsy), and prognosis in myocarditis. The objective of this multicenter, prospective, randomized, double-blind placebo-controlled trial is to assess the efficacy and safety of 12 - month treatment with prednisone and azathioprine comparing to placebo on top of guideline-recommended medical therapy in patients with biopsy-proven virus negative myocarditis or inflammatory cardiomyopathy and reduced ejection fraction (LVEF ≤ 45%). The study will also assess persistence of the treatment effects after 12 months.

DETAILED DESCRIPTION:
Myocarditis/ inflammatory cardiomyopathy, which often leads to heart failure (HF), is still an under-studied disease with various clinical manifestations. The active myocarditis is found post-mortem even in 42% of sudden deaths of young people and in 9-16% of adults and 46% of children with idiopathic dilated cardiomyopathy. Moreover, an increase in morbidity and mortality from myocarditis was recorded in the years 1990-2015. Myocarditis significantly increases the risk of HF, serious arrhythmias and conduction abnormalities, sudden death, anxiety, depression and it reduces quality of life. Myocarditis affects mainly young people (18-40 years old, and children) who lead active family life and work. Therefore, the disease causes deterioration of entire family life, it reduces individual productivity, creates high and long-term treatment costs. There is an urgent need to improve myocarditis therapy. Current guidelines recommendations in myocarditis consists of standard treatment of already developed HF and long-term avoidance of physical activity. Due to the lack of good quality scientific data, there is no clear recommendation for the targeted treatment - thus patients' prognosis may be poor. The pathogenesis of myocarditis and limited reports suggest the reasonable chance of significant improvement of patients' survival due to immunosuppressive therapy.

Aim: Aim of the IMPROVE-MC study is to assess the efficacy and safety of 12-month immunosuppressive treatment with prednisone and azathioprine compared with placebo on the guideline-recommended medical therapy in patients with biopsy-proven virus-negative myocarditis or inflammatory cardiomyopathy. Secondary aim is to create ready-to-use diagnostic and therapeutic scheme in polish and international healthcare systems, which can lead to myocarditis guidelines change.

Population and methods: In this multicenter (7 recruitment centers), prospective, randomized, double-blind placebo-controlled trial we are going to include 100 patients aged 18-65 years old, with biopsy-proven virus-negative myocarditis in stable or worsening course of the disease despite standard medical treatment, with left ventricular ejection fraction (LVEF) ≤45% and/or significant cardiac arrhythmias refractory to antiarrhythmic treatment.

Exclusion criteria consist of ie.: another specific etiology of HF different from myocarditis; already implanted ventricular assist device; a heart transplant recipient; contraindications to immunosuppressive treatment; suspected sarcoidosis or giant cell myocarditis.

Intervention: azathioprine for 12 months and prednisone for the first 6 months versus placebo for 12 months Study course: after randomization patients will undergo one-year double-blind treatment and then one-year follow-up to assess the long-term effects of the treatment.

The efficacy and safety of the treatment will be assessed during study visits: investigational products/ placebo will be provided and additional tests will be performed - 48-hour Holter monitoring, echocardiography, cardiac magnetic resonance imaging (CMR), laboratory tests and follow-up endomyocardial biopsy (EMB) after one-year of treatment. In order to broaden knowledge about myocarditis pathogenesis additional genetic, immunology and proteomic tests will be performed. All echo, MRI, Holter and biopsy tests will be evaluated centrally.

Study endpoints:

primary endpoint is LVEF at 12-months. secondary endpoints include analysis of: e.g. clinical outcomes, echocardiography, CMR, EMB, laboratory examinations, quality of life and heart failure questionnaires.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in this study, patient must fulfill all of the following inclusion criteria:

1. Written informed consent to participate in the IMPROVE-MC study (including two EMBs and two cardiac CMRs) prior to any evaluation or procedure related to the study.
2. Patient with clinically suspected myocarditis or inflammatory cardiomyopathy (according to the criteria of the ESC Working Group on Myocardial & Pericardial Diseases 2013 and ESC Heart Failure Guidelines 2021); OR/ AND, Patients with already diagnosed active myocarditis (lymphocytic or eosinophilic) or inflammatory cardiomyopathy who will undergo diagnostic right ventricular (or/and left ventricular) EMB during the screening; OR / AND, Patients with already diagnosed active myocarditis (lymphocytic or eosinophilic) or inflammatory cardiomyopathy confirmed by right ventricular (or/and left ventricular) EMB that was performed according to the IMPROVE-MC study protocol within 3 months from screening.
3. Men or women aged 18-65. Women of childbearing age must have a negative pregnancy test result. Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (with a failure rate of < 1% per year) for the duration of the study (from the time they sign consent) and for 8 weeks after the last dose of study treatment to prevent pregnancy. Patients agreeing to total sexual abstinence can also be included, assuming it is their usual lifestyle. Women are considered postmenopausal and without the potential to have a child if they have 12 months of natural (spontaneous) amenorrhea with an appropriate clinical picture (e.g. appropriate age, history of vasomotor symptoms) or have undergone bilateral surgical ovariectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of ovariectomy alone, only if the reproductive status of the woman has been confirmed by assessing hormone levels.
4. No significant improvement in clinical condition or worsening course of the disease despite the standard treatment in the investigator's opinion, in the last ≥ 3 months prior to the screening period.
5. LVEF 10 - 45% measured by echocardiogram taken during the screening period

   1. No significant LVEF improvement in the last ≥3 months prior to the screening period in the investigator's opinion.
   2. LVEF should be measured under stable conditions as assessed by the investigator.
   3. LVEF should be verified in the CORE-LAB.
6. Histological and immunohistochemical evidence of active myocarditis (lymphocytic or eosinophilic) OR inflammatory cardiomyopathy during the screening period (EMB during the screening or within last 3 months).
7. Absence of cardiotropic viruses in cardiac tissue at PCR analysis during the screening period (EMB during the screening or within last 3 months).

Exclusion Criteria:

Patients fulfilling any of the following exclusion criteria are not eligible for inclusion in this study. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

1. Presence of contraindications to immunosuppressive therapy with steroids and/ or azathioprine (including hypersensitivity to azathioprine/ 6-mercaptopurine or prednisone, mainly untreated systemic infection, uncontrolled diabetes, poorly controlled endocrine diseases, osteoporosis, active gastric or duodenal ulcer, uncontrolled hypertension, leukocytopenia (leukocyte counts <4 x 109/l), neutropenia (neutrophils <1.5 x 109/l), thrombocytopenia (platelet levels <130 x 109/l), anemia (hemoglobin levels <11 g/dl).
2. Positive clinical screening for active infections, including HIV, HBV, HCV. Assessment of tuberculosis infection should be considered before screening, according to the local epidemiologic status and according to investigator's opinion. After careful evaluation of the activity of the infection (or cure of the infection), the patient may continue participation in the study according to investigator's opinion.
3. Another specific cause of heart failure (including severe congenital, valvular, hypertensive, and/or coronary artery disease) that could justify the severity of cardiac dysfunction.
4. Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), storage diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, genetic hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy or known pericardial constriction.
5. Diagnosed or suspected cardiac sarcoidosis or giant cell myocarditis, autoimmune/ systemic immune-mediated disease (i.e. granulomatosis with polyangiitis, lupus erythematosus) that might require specific immunosuppressive therapy. Recent, current or expected future need for long-term use of immunosuppressive therapy with steroids and/ or azathioprine and/ or other immunosuppressive agent (caution - short-term course of steroids [i.e. for asthma attack, occasional topical applications] is not an exclusion).
6. NYHA class I and IV.
7. Subjects with body mass index >40 kg/m2 or body weight <50 kg.
8. Pregnancy, lactation or women who plan to become pregnant during the trial. Lack of consent to the use of effective forms of contraception.
9. Any documented or suspected active malignant neoplasm or history of malignant neoplasm within the 5 years prior to the screening period.
10. History of cytostatic therapy or radiotherapy.
11. Liver disease defined as any of the following: AST or ALT or ALP above 3x ULN; bilirubin >1.5 mg/dL.
12. Impaired renal function, defined as eGFR <45 mL / min / 1.73 m2 (CKD-EPI) measured under stable condition or requiring dialysis. Conditionally, according to the investigator's decision, patients with eGFR 40-45 ml / min / 1.73 m2 may be included.
13. The need or refusal to stop taking any drug considered to interfere with the safe course of the study (e.g., allopurinol).
14. Currently implanted or planned VAD, CRT or heart transplant.
15. Patients with pacemaker or ICD requiring a high percentage of ventricular pacing (>30%) which could influence the result of LVEF measurement in the investigator's opinion.
16. Gastrointestinal surgery or gastrointestinal disorder that could interfere with trial drug(s) absorption in the investigator's opinion.
17. History or presence of any other disease with a life expectancy <3 years.
18. Any contraindications or intolerance to CMR*, including but not limited to:

    1. the presence of cardiac implantable electronic device implanted <6 weeks ago;
    2. pacing capture threshold out of the normal range;
    3. additional cardiac leads (particularly abandoned pacemaker leads), epicardial leads, fractured leads, additional components such as lead adapters or lead extension;
    4. aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body that could be contraindication to CMR;
    5. presence of claustrophobia making impossible to perform CMR;
    6. or any other clinical history or study that determines that, in the investigator's judgment, the performance of an CMR may pose a potential risk to the patient.
19. Immunization with live organism vaccines in the last 3 months prior to randomization.
20. Chronic alcohol or drug abuse or non-compliance with medical recommendations or any condition that, in the investigator's opinion, makes patient an unreliable trial subject or unlikely to complete the trial.
21. Use of other investigational drugs at the time of enrollment, or within 30 days, or within 5 half-lives of enrollment, whichever is longer.
22. Subjects directly involved in the execution of this protocol.

    * CMR in non-conditional CIED proved to be safe. CMR in CIED patients will be performed according to HRS 2017 and ESC Pacing 2021 guidelines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
LVEF at 12 - months. | 12- months
  Left ventricle ejection fraction (LVEF) at 12 - months.

SECONDARY OUTCOMES:
Proportion of patients who responded to immunosuppressive therapy. | 12-months
  Proportion of patients who responded to immunosuppressive therapy as defined by an LVEF increase of ≥10% over time.
LVEF at 12 months in subgroups of patients with baseline LVEF ≤30% and >30% | 12 months
Change in the LV end-systolic and end-diastolic dimensions as well as the LV end-systolic and end-diastolic volumes over time. | 12-months
Change from baseline in NYHA class over time. | 12-months
Occurrence of adjudicated heart failure decompensation (hospitalization or ambulatory visit). | 12-months
Change from baseline in percentage of patients in NYHA III/IV and NYHA II class over time. | assessed up to 24th month from the randomization
  Change from baseline in percentage of patients in NYHA III/IV and NYHA II class over time (compared to baseline and to the end of treatment)
Occurrence of need for diuretic i.v. administration. | assessed up to 24th month from the randomization
Change from baseline in 6 minute walk test (6MWT) distance over time. | assessed up to 24th month from the randomization
Time to first adjudicated hospitalization for heart failure. | assessed up to 24th month from the randomization
Time to first all-cause hospitalization. | assessed up to 24th month from the randomization
Occurrence (first and recurrent) of all-cause hospitalization, heart failure hospitalization, heart failure outpatient visit, myocarditis or inflammatory cardiomyopathy recurrence, all-cause death, heart transplantation, implantation of cardiac device | assessed up to 24th month from the randomization
  Occurrence (first and recurrent) of all-cause hospitalization, heart failure hospitalization, heart failure outpatient visit, myocarditis or inflammatory cardiomyopathy recurrence, all-cause death, heart transplantation, implantation of cardiac device (pacemaker, implantable cardioverter-defibrillator, cardiac resynchronization therapy, ventricular assist device) assessed in combination or independently.
New onset atrial fibrillation (AF). | assessed up to 24th month from the randomization
New onset sustained ventricular tachycardia (VT) or ventricular fibrillation (VF). | assessed up to 24th month from the randomization
≥50% reduction from baseline in ventricular ectopic beats (VEBs) number in 48h Holter monitoring over time. | assessed up to 24th month from the randomization
≥50% reduction from baseline in nonsustained VT number in 48h Holter monitoring over time. | assessed up to 24th month from the randomization
≥50% reduction from baseline in AF burden in 48h Holter monitoring over time. | assessed up to 24th month from the randomization
Changes from baseline in CMR results | assessed up to 24th month from the randomization
  Changes from baseline in CMR results (early gadolinum enhancement (EGE), late gadolinum enhancement (LGE), edema, LV dimensions and volumes, T1/T2 mapping) after one-year.
Changes from baseline in concentration of biomarkers of fibrosis and myocardial necrosis (troponin I, NT-proBNP, sST2, Gal-3) over time. | assessed up to 24th month from the randomization
Qualitative and quantitative change from baseline in inflammatory infiltration, human leukocyte antigen (HLA) expression and fibrosis in EMB after one-year. | after 12- months
Change from baseline in KCCQ (Kansas City Cardiomyopathy Questionnaire) overall summary score over time. | assessed up to 24th month from the randomization
Change from baseline in KCCQ (Kansas City Cardiomyopathy Questionnaire) total symptom score over time. | assessed up to 24th month from the randomization
Change from baseline in KCCQ (Kansas City Cardiomyopathy Questionnaire) individual domains over time. | assessed up to 24th month from the randomization
Change from baseline in KCCQ (Kansas City Cardiomyopathy Questionnaire) based on patient-preferred outcome over time. | assessed up to 24th month from the randomization
Change from baseline in SF-36 (36-Item Short Form Survey) questionnaire overall summary score over time. | assessed up to 24th month from the randomization
Change from baseline in PGI-I (Patients Global Impression of Improvement) scale over time. | assessed up to 24th month from the randomization
Change from baseline in CGI-I (Clinical Global Impressions - Improvement) scale over time. | assessed up to 24th month from the randomization
Change from baseline in health economic analysis by HCRU (Healthcare Resource Utilization). | assessed up to 24th month from the randomization
Occurrence of need for inotropic drugs/nitroglycerin i.v. administration | assessed up to 24th month from the randomization
  Occurrence of need for inotropic drugs/nitroglycerin i.v. administration
LVEF at 24 months | compared to baseline and/or to the end of treatment) analyzed during follow up (13-24 months)
  LVEF at 24 months (maintenance or further improvement).
LVEF at 24 months in subgroups of patients with baseline LVEF ≤30% and >30% | compared to baseline and/or to the end of treatment) analyzed during follow up (13-24 months)
  LVEF at 24 months (maintenance or further improvement) in subgroups of patients with baseline LVEF ≤30% and >30%
Change in the LV end-systolic and end-diastolic dimensions as well as the LV end-systolic and end-diastolic volumes over time. | compared to baseline and/or to the end of treatment) analyzed during follow up (13-24 months)
Change in NYHA class over time | compared to baseline and/or to the end of treatment) analyzed during follow up (13-24 months)
Occurrence of adjudicated heart failure decompensation (hospitalization or ambulatory visit). | analyzed during follow up (13-24 months)
Application of mechanical circulatory support (i.e. ECMO). | assessed up to 24th month from the randomization
≥50% increase from the end of treatment in VEBs number in 48h Holter monitoring over time. | assessed from the end of treatment up to 24th months from the randomization
≥50% increase from the end of treatment in nonsustained VT number in 48h Holter monitoring over time | assessed from the end of treatment up to 24th months from the randomization
≥50% increase from the end of treatment in AF burden in 48h Holter monitoring over time | assessed from the end of treatment up to 24th months from the randomization
Changes in tricuspid annular plane systolic excursion | assessed up to 24th months from the randomization
  Changes in tricuspid annular plane systolic excursion (reported in centimeters) over time.
Changes in dimensions of the heart cavities | assessed up to 24th months from the randomization
  Changes in dimensions of the heart cavities (ventricles and atria; reported in centimeters) over time.
Changes in volumes of the heart cavities | assessed up to 24th months from the randomization
  Changes in volumes of the heart cavities (ventricles and atria; reported in milliliters) over time.
Changes in thickness of left and right ventricles | assessed up to 24th months from the randomization
  Changes in thickness of left and right ventricles (reported in centimeters) over time.
Changes in tissue Doppler velocities (medial and lateral) of the mitral annulus | assessed up to 24th months from the randomization
  Tissue Doppler velocities (medial and lateral) of the mitral annulus (reported in centimeters per second) over time.
Changes in strain of heart cavities | assessed up to 24th months from the randomization
  Changes in strain of heart cavities (ventricles and atria; reported as a percentage) over time.
Changes in concentration of biomarkers of fibrosis and myocardial necrosis (troponin I, NT-proBNP) over time | assessed up to 24th months from the randomization
Changes in concentration of anti-heart autoantibodies (AHA) over time | assessed up to 24th months from the randomization
Change of patients' health status as assessed by the patients self-reported EQ-5D over time. | assessed up to 24th months from the randomization
Change in clinical summary score (heart failure symptoms and physical limitations domains) of KCCQ Questionnaire over time | assessed up to 24th months from the randomization
Cost-effectiveness analysis | assessed up to 24th months from the randomization
  Pharmacoeconomic analysis based on questionnaires (SF-36, KCCQ, EQ-5D-5L, PGI, CGI, HCRU) and patient prognosis (including adverse event rates, hospitalizations, death, worsening of heart failure, arrhythmias, drug-related adverse events, change in LVEF and NYHA class, gain of QALY).

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Grabowski, Professor, Study Chair — Medical University of Warsaw; Krzysztof Ozierański, MD, PhD, Principal Investigator — Medical University of Warsaw; Agata Tymińska, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- First Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
the study documents will be available on demand
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the study completion
Access Criteria: On demand